CLINICAL TRIAL: NCT03591549
Title: Role of Fulvestrant in The Treatment of Metastatic Breast Cancer in Premenopausal Women
Brief Title: Fulvestrant in Metastatic Breast Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AIMekkawy, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RFTMBCPW
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Goserelin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fulvestrant arm (Experimental): patients will receive fulvestrant + zoladex intramuscular monthly with an assessment every three months to assess the response and progression
  Interventions: Drug: Faslodex; Drug: Zoladex

INTERVENTIONS:
Drug: Faslodex — intramuscular injection monthly
Drug: Zoladex — intramuscular injection monthly

SUMMARY:
This is a prospective study of the role of fulvestrant in combination with ovarian function suppression as first-line therapy in premenopausal patients with metastatic hormone receptor-positive breast cancer.

DETAILED DESCRIPTION:
Hormone receptor-positive breast cancer is the most common presentation of breast cancer today. Endocrine therapy is the preferred treatment modality in hormone receptor-positive early stage and advanced breast cancer.

Fulvestrant is an estrogen receptor antagonist indicated for the treatment of postmenopausal women with estrogen receptor-positive, locally advanced or metastatic breast cancer for disease relapse on or after adjuvant antiestrogen therapy, or disease progression on therapy with an antiestrogen.

Fulvestrant is a selective estrogen receptor down-regulator that competitively binds to estrogen receptors, with a binding affinity approximately 100 times greater than that of tamoxifen. Once bound to the receptor, estrogen receptor dimerization and nuclear translocation are inhibited, resulting in accelerated receptor degradation. Besides the nuclear estrogen receptor, fulvestrant blocks cytoplasmatic as well as membrane-bound receptors. It is therefore suggested that fulvestrant inhibits the estrogen receptor/growth factor crosstalk responsible for estrogen receptor activation in the absence of estrogen.

In premenopausal women, the combination of gonadotropin-releasing hormone analogues and tamoxifen is a standard of care for premenopausal women with endocrine-responsive metastatic breast cancer. Upon disease progression, selected patients may be candidates for further endocrine treatment in combination with ongoing ovarian function suppression.

Several preclinical studies have demonstrated that fulvestrant was markedly more effective than tamoxifen in inhibiting the in vitro growth of human breast carcinoma cells and was also effective in tamoxifen-resistant breast carcinoma xenografts in vivo mouse models.

Fulvestrant has also been shown to be active in patients previously untreated with endocrine therapies, either in the neoadjuvant or in the metastatic setting, alone or in combination with other therapies such as AI or targeted drugs.

In a study done by Bartsch R et al revealed that complete response was observed in a single patient, partial response in three and disease stabilization ≥ 6 months in eleven patients, resulting in a CBR of 58%. Median time to progression was 6 months and overall survival 32 months in premenopausal women treated by fulvestrant for metastatic breast cancer.

The efficacy of fulvestrant, a selective estrogen receptor degrader, has been demonstrated in hormone receptor-positive breast cancer patients previously untreated or treated with hormonal therapy. In a phase III trials, fulvestrant has demonstrated equivalent or improved clinical efficacy when compared with established endocrine agents. Presently, fulvestrant is licensed globally as first-line endocrine management for advanced breast cancer in post-menopausal women.

In the metastatic setting of premenopausal breast cancer, tamoxifen or aromatase inhibitors, both with ovarian suppression/ablation, should be the preferred choice, unless rapid tumor shrinkage is needed. No data are available with fulvestrant in young patients.

Fulvestrant received a new Food Drug Administration indication in December 2016, in combination with palbociclib, both in pre/peri/postmenopausal women with breast cancer progressing after endocrine therapy.

Regarding the optimal dose of fulvestrant, the FIRST trial indicated superior efficacy of fulvestrant 500 mg, therefore fulvestrant in premenopausal women should be used in high-dose/loading-dose regimen.

Main toxicity of the fulvestrant that reported was vasomotor symptoms (hot flushes) and gastrointestinal side-effects such as nausea, vomiting, anorexia, diarrhea and abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

* Women with age 30-50 years old (premenopause).
* Histological confirmation of metastatic disease.
* Hormonal receptor positive.
* Endocrine therapy for early disease had been completed more than 12 months before the study (patients who was not resistance to hormonal therapy).
* Metastatic breast cancer at presentation.
* Patients had not received any previous systemic therapy for metastatic disease.
* Performance status (ECOG) 0-2.

Exclusion Criteria:

* Patient >55 years old.
* Non-histologically diagnosed.
* Hormonal receptor negative
* Non metastatic
* received previous line therapy in the metastatic setting.
* Patient with performance >2.
* Patient with co-morbidity
* Patients with brain metastasis

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 30 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | three years
  time from start of the treatment till progression of the disease

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bartsch R, Bago-Horvath Z, Berghoff A, DeVries C, Pluschnig U, Dubsky P, Rudas M, Mader RM, Rottenfusser A, Fitzal F, Gnant M, Zielinski CC, Steger GG. Ovarian function suppression and fulvestrant as endocrine therapy in premenopausal women with metastatic breast cancer. Eur J Cancer. 2012 Sep;48(13):1932-8. doi: 10.1016/j.ejca.2012.03.002. Epub 2012 Mar 27. PMID 22459763
- [Background] Wakeling AE, Dukes M, Bowler J. A potent specific pure antiestrogen with clinical potential. Cancer Res. 1991 Aug 1;51(15):3867-73. PMID 1855205
- [Background] Fawell SE, White R, Hoare S, Sydenham M, Page M, Parker MG. Inhibition of estrogen receptor-DNA binding by the "pure" antiestrogen ICI 164,384 appears to be mediated by impaired receptor dimerization. Proc Natl Acad Sci U S A. 1990 Sep;87(17):6883-7. doi: 10.1073/pnas.87.17.6883. PMID 2395882
- [Background] Wakeling AE. Similarities and distinctions in the mode of action of different classes of antioestrogens. Endocr Relat Cancer. 2000 Mar;7(1):17-28. doi: 10.1677/erc.0.0070017. No abstract available. PMID 10808193